CLINICAL TRIAL: NCT03694756
Title: TMEM-MRI: A Pilot Feasibility Study of Magnetic Resonance Imaging for Imaging of TMEM (Tumor Microenvironment of Metastasis) in Patients With Operable Breast Cancer
Brief Title: TMEM-MRI: A Pilot Feasibility Study of MRI for Imaging of TMEM in Patients With Operable Breast Cancer
Acronym: TMEM-MRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-9529
Record Dates: First submitted 2018-09-28; First posted 2018-10-03 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: TMEM;; Magnetic resonance imaging (MRI)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients were originally intended to be enrolled in 2 cohorts (A and B), based on breast biopsy status; however, the study design was changed following Protocol Amendment.
Masking Description: No need for masking, all patients will undergo TMEM-MRI
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Pre-biopsy patients (Cohort A) (Other): Patients identified by radiologist at the time of diagnostic evaluation and TMEM-MRI scheduled. After TMEM-MRI, the patient will undergo core biopsy as per usual radiology procedure, with additional fine-needle aspiration (FNA) preceding the core biopsy). After the breast biopsy confirms the suspected diagnosis of invasive breast carcinoma, the patient will be referred to breast surgery and a treatment plan devised per National Comprehensive Cancer Network/American Society of Clinical Oncology (NCCN/ASCO) guidelines.
  No patients were enrolled into this arm/group and Cohort A has been removed by protocol amendment. This was intended to be a cohort for patients before breast biopsy in the event the biopsy procedure created a hematoma which would, in turn, affect measurement of TMEM-MRI activity. Since this effect was not observed in the first set of patients enrolled, Cohort A was removed from the study and only patients post-breast biopsy were enrolled (Cohort B).
  Interventions: Device: TMEM-MRI; Procedure: FNA
- Post-biopsy patients (Cohort B) (Other): Patients after breast biopsy. Once consent is obtained, patients will undergo TMEM-MRI. The patients will undergo definitive breast surgery and will receive adjuvant treatments as per NCCN/ASCO guidelines. TMEM density, MenaCalc and MenaINV will be evaluated in final surgical specimen. Uth qTPERM will be correlated with TMEM density, MenaCalc and MenaINV.
  Interventions: Device: TMEM-MRI
- Post-neoadjuvant therapy patients (Cohort C) (Other): Patients status post neoadjuvant therapy. Patients who received neoadjuvant will be enrolled into Cohort C to understand the correlation between TMEM MRI activity and TMEM doorway density following after neoadjuvant chemotherapy. Only patients with residual palpable mass on physical exam will be included (≥ 1cm). Patients will undergo TMEM-MRI after neoadjuvant therapy is completed. Patients will also have CTCs and circulating tumor DNA (ctDNA) measured on the same day of TMEM-MRI (+/- 3 days). TMEM density, MenaCalc and MenaINV will be evaluated in breast surgical specimen (after pre-operative therapy). Uth qTPERM will be correlated with TMEM density, MenaCalc and MenaINV after pre-operative therapy.
  Interventions: Device: TMEM-MRI

INTERVENTIONS:
Device: TMEM-MRI — TMEM MRI INFORMATION: Unilateral breast MRI will be obtained on a 3.0T whole body MRI scanner with a dedicated breast radiofrequency coil. The patient will be scanned in the prone position with an in-dwelling IV catheter for a single dose contrast agent injection.
Procedure: FNA — FNA: The patients who are recruited prior to biopsy (Cohort A) will have had TMEM-MRI performed prior to biopsy. They will then present to radiology for ultrasound-guided core biopsy of the breast mass. FNA will be performed during this procedure. The FNA will be performed after local anesthetic is administered but prior to insertion of the core biopsy needle. FNA will be performed by the radiologist under direct sonographic visualization of the mass. Five passes will be obtained with a 25-gauge needle. The FNA material will be expelled into 1.5 ml Eppendorf tube containing phosphate buffered saline with Ethylenediaminetetraacetic acid (EDTA).
  Arms: Pre-biopsy patients (Cohort A)

SUMMARY:
The aim of this study is to assess feasibility of a new imaging technology in the management of breast cancer - Tumor Microenvironment of Metastasis - Magnetic Resonance imaging (TMEM-MRI).

DETAILED DESCRIPTION:
The primary objective of this study is to develop a magnetic resonance imaging (MRI) based method for assessing TMEM-mediated permeability associated with cancer cell dissemination in breast cancer patients. TMEM-MRI has the ability to detect tumor areas with more leakiness (perfusion), where cancer cells enter blood vessels to travel to other sites. This novel TMEM-MRI has potential to be used in clinical practice to identify tumors with high leakiness that might have higher chances to recur after breast cancer treatment. In addition, TMEM-MRI can potentially be used to assess response to preoperative treatments (chemotherapy, hormonal therapy) over time.

In a prior study, it was found that patients with high TMEM doorway score, compared to patients with mid/low TMEM doorway score, in their residual disease after neoadjuvant therapy, had worse distant relapse-free survival (p = 0.008). These results demonstrated that TMEM doorway density after neoadjuvant therapy is a prognostic biomarker of breast cancer outcomes. In the initial development of the proposed TMEM MRI in humans, the tumor microenvironment is naïve to treatment. However, neoadjuvant therapy may affect the tumor microenvironment which could affect vascular anatomy - a key component of the TMEM MRI algorithm. Therefore, the study team aims to assess the correlation between TMEM doorway density and TMEM MRI activity after neoadjuvant therapy (Pilot Cohort C).

ELIGIBILITY:
Inclusion Criteria

* For pre-pilot phase (MRI sequence development):

  o Patients with a breast mass, with biopsy-proven histology of invasive breast carcinoma (any histologic type and ER,PR,HER2 status)
* For pilot phase Cohort A:

  o Patients with a breast mass considered highly suspicious for invasive carcinoma by the radiologist (BIRADS 5).
* For pilot phase Cohort B:

  * Patients with a breast mass found to be invasive ductal carcinoma on core biopsy.
  * No preoperative therapy for the current breast cancer has been started (endocrine therapy, chemotherapy, or radiation). Patients can receive preoperative treatment after TMEM-MRI is conducted, if clinically indicated.
* For pilot phase Cohort C:

  * Patients with locally advanced breast cancer, anatomic stage II-III, who received neoadjuvant therapy as per standard of care.
  * Residual palpable mass > 1 cm in largest diameter after neoadjuvant therapy.
  * Candidate for breast MRI before definitive surgery.
* Tumor size/breast mass should be > 1 cm in largest diameter (radiologically).
* Multifocal disease is allowed, as long as patients meet all eligibility criteria.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Willingness to undergo a "research breast MRI".
* Patient must be able to undergo MRI with gadolinium enhancement.

  * No history of untreatable claustrophobia.
  * No presence of non-MRI compatible metallic objects or metallic objects that, in the opinion of a radiologist, would make MRI a contraindication.
  * No history of sickle cell disease.
  * No contraindication to intravenous contrast administration.
  * No known allergy-like reaction to gadolinium
  * No known or suspected renal impairment. Glomerular Filtration Rate (GFR) should be greater than 30 mL/min/1.73 m2.
* Weight less than or equal to the MRI table limit.
* Ability to understand and willingness to sign a written informed consent.

Exclusion Criteria

* Patients may not have had breast cancer or radiation therapy to the ipsilateral breast in the past.
* No breast prosthetic implants (silicone or saline) are allowed.
* Use of any investigational agent within 30 days of starting study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study.
* Patients must be non-pregnant and non-lactating. Patients must have a negative pregnancy test (urine or serum) within 7 days of registration date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Tumor permeability assessed by TMEM-MRI | Cohort B: ~14 days following breast biopsy and signing of consent. Cohort C: After neoadjuvant therapy and signing of consent and 0-56 days before surgery
  Tumor permeability will be assessed by TMEM-MRI, and is defined as a number of Uth units (the number of tumor voxels with permeability density above threshold divided by the number of all tumor voxels) that will be obtained from the permeability map and TMEM-MRI algorithm.

SECONDARY OUTCOMES:
TMEM density in breast cancer patients | Cohort B: ~14 days following breast biopsy and consent. Cohort C: After neoadjuvant therapy and signing of consent analyses. Conducted on tissue sections from formalin-fixed paraffin-embedded breast cancer specimen resected for therapeutic purposes
  TMEM density is defined as the number of TMEM units visualized by triple immunohistochemistry in 10 high power fields (40X). TMEM density will be measured with a fully automated and scalable clinical assay for identification and enumeration of TMEM utilizing digital pathology methods coupled with image analysis
MenaCalc | Cohort B: ~14 days following breast biopsy and consent. Cohort C: After neoadjuvant therapy and signing of consent analyses. Conducted on tissue sections from formalin-fixed paraffin-embedded breast cancer specimen resected for therapeutic purposes
  MenaCalc is calculated by subtracting the Z-score value of Mena11a from the Z-score value of pan-Mena, obtained by quantitative immunohistochemistry in formalin-fixed paraffin-embedded breast tumor specimens. MenaCalc can also be measured by quantitative reverse transcription polymerase chain reaction (qRT-PCR) in cancer cells obtained by FNA
MenaInv | Cohort B: ~14 days following breast biopsy and consent. Cohort C: After neoadjuvant therapy and signing of consent analyses. Conducted on tissue sections from formalin-fixed paraffin-embedded breast cancer specimen resected for therapeutic purposes
  MenaInv is calculated as pixel intensity obtained by quantitative immunofluorescence per area of formalin-fixed paraffin-embedded tumor tissue. MenaINV can also be measured by qRT-PCR in cancer cells obtained by FNA
Circulating Tumor Cells (CTCs) | Cohort B: ~14 days following breast biopsy and signing of consent. Cohort C: After neoadjuvant therapy and consent and 0-56 days before surgery
  CTCs will detected and enumerated from peripheral blood samples using EPIC sciences or RareCyte platform. Patients will undergo venipuncture to obtain specimen for CTC assays. Specimens will be shipped to EPIC sciences (using CTC liquid biopsy blood collection kit) or the University of Southern California (using RareCyte collection kit) to be processed and analyzed as per respective protocols. CTCs will be measured +/- 3 days of TMEM-MRI. Group mean results in number of cells/mL of peripheral blood will be reported for patients in pilot phase Cohort B and pilot phase Cohort C.

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Anampa, MD, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Hellman, S. and J.R. Harris, Natural history of breast cancer, in Diseases of the Breast., J.R. eds Harris, Lippman, M. E., Morrow, M. & Osborne, C. K., Editor. 2000, Lippincott Williams & Wilkins: Philadelphia. p. 407-23.
- [Background] Weigelt B, Peterse JL, van 't Veer LJ. Breast cancer metastasis: markers and models. Nat Rev Cancer. 2005 Aug;5(8):591-602. doi: 10.1038/nrc1670. PMID 16056258
- [Background] Thiery JP, Acloque H, Huang RY, Nieto MA. Epithelial-mesenchymal transitions in development and disease. Cell. 2009 Nov 25;139(5):871-90. doi: 10.1016/j.cell.2009.11.007. PMID 19945376
- [Background] Fidler IJ, Poste G. The "seed and soil" hypothesis revisited. Lancet Oncol. 2008 Aug;9(8):808. doi: 10.1016/S1470-2045(08)70201-8. No abstract available. PMID 18672217
- [Background] Kalluri R, Weinberg RA. The basics of epithelial-mesenchymal transition. J Clin Invest. 2009 Jun;119(6):1420-8. doi: 10.1172/JCI39104. PMID 19487818
- [Background] Warzecha CC, Carstens RP. Complex changes in alternative pre-mRNA splicing play a central role in the epithelial-to-mesenchymal transition (EMT). Semin Cancer Biol. 2012 Oct;22(5-6):417-27. doi: 10.1016/j.semcancer.2012.04.003. Epub 2012 Apr 23. PMID 22548723
- [Background] Ellis JD, Barrios-Rodiles M, Colak R, Irimia M, Kim T, Calarco JA, Wang X, Pan Q, O'Hanlon D, Kim PM, Wrana JL, Blencowe BJ. Tissue-specific alternative splicing remodels protein-protein interaction networks. Mol Cell. 2012 Jun 29;46(6):884-92. doi: 10.1016/j.molcel.2012.05.037. PMID 22749401
- [Background] Gertler F, Condeelis J. Metastasis: tumor cells becoming MENAcing. Trends Cell Biol. 2011 Feb;21(2):81-90. doi: 10.1016/j.tcb.2010.10.001. Epub 2010 Nov 9. PMID 21071226
- [Background] Shapiro IM, Cheng AW, Flytzanis NC, Balsamo M, Condeelis JS, Oktay MH, Burge CB, Gertler FB. An EMT-driven alternative splicing program occurs in human breast cancer and modulates cellular phenotype. PLoS Genet. 2011 Aug;7(8):e1002218. doi: 10.1371/journal.pgen.1002218. Epub 2011 Aug 18. PMID 21876675
- [Background] Agarwal S, Gertler FB, Balsamo M, Condeelis JS, Camp RL, Xue X, Lin J, Rohan TE, Rimm DL. Quantitative assessment of invasive mena isoforms (Menacalc) as an independent prognostic marker in breast cancer. Breast Cancer Res. 2012 Sep 12;14(5):R124. doi: 10.1186/bcr3318. PMID 22971274
- [Background] Forse CL, Agarwal S, Pinnaduwage D, Gertler F, Condeelis JS, Lin J, Xue X, Johung K, Mulligan AM, Rohan TE, Bull SB, Andrulis IL. Menacalc, a quantitative method of metastasis assessment, as a prognostic marker for axillary node-negative breast cancer. BMC Cancer. 2015 Jun 27;15:483. doi: 10.1186/s12885-015-1468-6. PMID 26112005
- [Background] Di Modugno F, Bronzi G, Scanlan MJ, Del Bello D, Cascioli S, Venturo I, Botti C, Nicotra MR, Mottolese M, Natali PG, Santoni A, Jager E, Nistico P. Human Mena protein, a serex-defined antigen overexpressed in breast cancer eliciting both humoral and CD8+ T-cell immune response. Int J Cancer. 2004 May 10;109(6):909-18. doi: 10.1002/ijc.20094. PMID 15027125
- [Background] Goswami S, Philippar U, Sun D, Patsialou A, Avraham J, Wang W, Di Modugno F, Nistico P, Gertler FB, Condeelis JS. Identification of invasion specific splice variants of the cytoskeletal protein Mena present in mammary tumor cells during invasion in vivo. Clin Exp Metastasis. 2009;26(2):153-9. doi: 10.1007/s10585-008-9225-8. Epub 2008 Nov 5. PMID 18985426
- [Background] Philippar U, Roussos ET, Oser M, Yamaguchi H, Kim HD, Giampieri S, Wang Y, Goswami S, Wyckoff JB, Lauffenburger DA, Sahai E, Condeelis JS, Gertler FB. A Mena invasion isoform potentiates EGF-induced carcinoma cell invasion and metastasis. Dev Cell. 2008 Dec;15(6):813-28. doi: 10.1016/j.devcel.2008.09.003. PMID 19081071
- [Background] Bear JE, Gertler FB. Ena/VASP: towards resolving a pointed controversy at the barbed end. J Cell Sci. 2009 Jun 15;122(Pt 12):1947-53. doi: 10.1242/jcs.038125. PMID 19494122
- [Background] Roussos ET, Balsamo M, Alford SK, Wyckoff JB, Gligorijevic B, Wang Y, Pozzuto M, Stobezki R, Goswami S, Segall JE, Lauffenburger DA, Bresnick AR, Gertler FB, Condeelis JS. Mena invasive (MenaINV) promotes multicellular streaming motility and transendothelial migration in a mouse model of breast cancer. J Cell Sci. 2011 Jul 1;124(Pt 13):2120-31. doi: 10.1242/jcs.086231. PMID 21670198
- [Background] Roussos ET, Goswami S, Balsamo M, Wang Y, Stobezki R, Adler E, Robinson BD, Jones JG, Gertler FB, Condeelis JS, Oktay MH. Mena invasive (Mena(INV)) and Mena11a isoforms play distinct roles in breast cancer cell cohesion and association with TMEM. Clin Exp Metastasis. 2011 Aug;28(6):515-27. doi: 10.1007/s10585-011-9388-6. Epub 2011 Apr 12. PMID 21484349
- [Background] Hughes SK, Oudin MJ, Tadros J, Neil J, Del Rosario A, Joughin BA, Ritsma L, Wyckoff J, Vasile E, Eddy R, Philippar U, Lussiez A, Condeelis JS, van Rheenen J, White F, Lauffenburger DA, Gertler FB. PTP1B-dependent regulation of receptor tyrosine kinase signaling by the actin-binding protein Mena. Mol Biol Cell. 2015 Nov 1;26(21):3867-78. doi: 10.1091/mbc.E15-06-0442. Epub 2015 Sep 2. PMID 26337385
- [Background] Weidmann MD, Surve CR, Eddy RJ, Chen X, Gertler FB, Sharma VP, Condeelis JS. MenaINV dysregulates cortactin phosphorylation to promote invadopodium maturation. Sci Rep. 2016 Nov 8;6:36142. doi: 10.1038/srep36142. PMID 27824079
- [Background] Pignatelli J, Goswami S, Jones JG, Rohan TE, Pieri E, Chen X, Adler E, Cox D, Maleki S, Bresnick A, Gertler FB, Condeelis JS, Oktay MH. Invasive breast carcinoma cells from patients exhibit MenaINV- and macrophage-dependent transendothelial migration. Sci Signal. 2014 Nov 25;7(353):ra112. doi: 10.1126/scisignal.2005329. PMID 25429076
- [Background] Patsialou A, Bravo-Cordero JJ, Wang Y, Entenberg D, Liu H, Clarke M, Condeelis JS. Intravital multiphoton imaging reveals multicellular streaming as a crucial component of in vivo cell migration in human breast tumors. Intravital. 2013 Apr 1;2(2):e25294. doi: 10.4161/intv.25294. PMID 25013744
- [Background] Roussos ET, Wang Y, Wyckoff JB, Sellers RS, Wang W, Li J, Pollard JW, Gertler FB, Condeelis JS. Mena deficiency delays tumor progression and decreases metastasis in polyoma middle-T transgenic mouse mammary tumors. Breast Cancer Res. 2010;12(6):R101. doi: 10.1186/bcr2784. Epub 2010 Nov 25. PMID 21108830
- [Background] Wyckoff J, Wang W, Lin EY, Wang Y, Pixley F, Stanley ER, Graf T, Pollard JW, Segall J, Condeelis J. A paracrine loop between tumor cells and macrophages is required for tumor cell migration in mammary tumors. Cancer Res. 2004 Oct 1;64(19):7022-9. doi: 10.1158/0008-5472.CAN-04-1449. PMID 15466195
- [Background] Wyckoff JB, Wang Y, Lin EY, Li JF, Goswami S, Stanley ER, Segall JE, Pollard JW, Condeelis J. Direct visualization of macrophage-assisted tumor cell intravasation in mammary tumors. Cancer Res. 2007 Mar 15;67(6):2649-56. doi: 10.1158/0008-5472.CAN-06-1823. PMID 17363585
- [Background] Falini B, Flenghi L, Pileri S, Gambacorta M, Bigerna B, Durkop H, Eitelbach F, Thiele J, Pacini R, Cavaliere A, et al. PG-M1: a new monoclonal antibody directed against a fixative-resistant epitope on the macrophage-restricted form of the CD68 molecule. Am J Pathol. 1993 May;142(5):1359-72. PMID 7684194
- [Background] Parums DV, Cordell JL, Micklem K, Heryet AR, Gatter KC, Mason DY. JC70: a new monoclonal antibody that detects vascular endothelium associated antigen on routinely processed tissue sections. J Clin Pathol. 1990 Sep;43(9):752-7. doi: 10.1136/jcp.43.9.752. PMID 2212067
- [Background] Robinson BD, Sica GL, Liu YF, Rohan TE, Gertler FB, Condeelis JS, Jones JG. Tumor microenvironment of metastasis in human breast carcinoma: a potential prognostic marker linked to hematogenous dissemination. Clin Cancer Res. 2009 Apr 1;15(7):2433-41. doi: 10.1158/1078-0432.CCR-08-2179. Epub 2009 Mar 24. PMID 19318480
- [Background] Rohan TE, Xue X, Lin HM, D'Alfonso TM, Ginter PS, Oktay MH, Robinson BD, Ginsberg M, Gertler FB, Glass AG, Sparano JA, Condeelis JS, Jones JG. Tumor microenvironment of metastasis and risk of distant metastasis of breast cancer. J Natl Cancer Inst. 2014 Jun 3;106(8):dju136. doi: 10.1093/jnci/dju136. Print 2014 Aug. PMID 24895374
- [Background] Dowsett M, Sestak I, Lopez-Knowles E, Sidhu K, Dunbier AK, Cowens JW, Ferree S, Storhoff J, Schaper C, Cuzick J. Comparison of PAM50 risk of recurrence score with oncotype DX and IHC4 for predicting risk of distant recurrence after endocrine therapy. J Clin Oncol. 2013 Aug 1;31(22):2783-90. doi: 10.1200/JCO.2012.46.1558. Epub 2013 Jul 1. PMID 23816962
- [Background] Sparano JA, Gray R, Oktay MH, Entenberg D, Rohan T, Xue X, Donovan M, Peterson M, Shuber A, Hamilton DA, D'Alfonso T, Goldstein LJ, Gertler F, Davidson NE, Condeelis J, Jones J. A metastasis biomarker (MetaSite Breast Score) is associated with distant recurrence in hormone receptor-positive, HER2-negative early-stage breast cancer. NPJ Breast Cancer. 2017 Nov 8;3:42. doi: 10.1038/s41523-017-0043-5. eCollection 2017. PMID 29138761
- [Background] Harney AS, Karagiannis GS, Pignatelli J, Smith BD, Kadioglu E, Wise SC, Hood MM, Kaufman MD, Leary CB, Lu WP, Al-Ani G, Chen X, Entenberg D, Oktay MH, Wang Y, Chun L, De Palma M, Jones JG, Flynn DL, Condeelis JS. The Selective Tie2 Inhibitor Rebastinib Blocks Recruitment and Function of Tie2Hi Macrophages in Breast Cancer and Pancreatic Neuroendocrine Tumors. Mol Cancer Ther. 2017 Nov;16(11):2486-2501. doi: 10.1158/1535-7163.MCT-17-0241. Epub 2017 Aug 24. PMID 28838996
- [Background] Kim G, Karadal-Ferrena B, Qin J, Sharma VP, Oktay IS, Lin Y, Ye X, Asiry S, Pastoriza JM, Cheng E, Ladak N, Condeelis JS, Adler E, Ginter PS, D'Alfonso T, Entenberg D, Xue X, Sparano JA, Oktay MH. Racial disparity in tumor microenvironment and distant recurrence in residual breast cancer after neoadjuvant chemotherapy. NPJ Breast Cancer. 2023 Jun 13;9(1):52. doi: 10.1038/s41523-023-00547-w. PMID 37311792
- [Background] Pignatelli J, Bravo-Cordero JJ, Roh-Johnson M, Gandhi SJ, Wang Y, Chen X, Eddy RJ, Xue A, Singer RH, Hodgson L, Oktay MH, Condeelis JS. Macrophage-dependent tumor cell transendothelial migration is mediated by Notch1/MenaINV-initiated invadopodium formation. Sci Rep. 2016 Nov 30;6:37874. doi: 10.1038/srep37874. PMID 27901093